CLINICAL TRIAL: NCT04315324
Title: A Phase I/II Study of AKR1C3-Activated Prodrug OBI-3424 (OBI-3424) In Patients With Relapsed/Refractory T-Cell Acute Lymphoblastic Leukemia (T-ALL)/T-Cell Lymphoblastic Lymphoma (T-LBL)
Brief Title: Study to Test OBI-3424 in Patients With T-Cell Acute Lymphoblastic Leukemia (T-ALL) or T-Cell Lymphoblastic Lymphoma (T-LBL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1905; NCI-2020-00768 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1905 (Other: SWOG); S1905 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Recurrent T Acute Lymphoblastic Leukemia; Refractory T Acute Lymphoblastic Leukemia; Refractory T Lymphoblastic Lymphoma; T Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Biopsy; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (AKR1C3-activated prodrug OBI-3424) (Experimental): Patients receive AKR1C3-activated prodrug OBI-3424 IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients who have not achieved a PR by the 4th cycle of treatment are removed from the study (unless clinically benefitting in the opinion of the treating investigator).Patients undergo blood sample collection during screening and CSF sample collection on study. Patients also undergo bone marrow aspirate or core biopsy and may undergo CT scan throughout the study.
  Interventions: Drug: AKR1C3-activated Prodrug AST-3424; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Computed Tomography

INTERVENTIONS:
Drug: AKR1C3-activated Prodrug AST-3424 — Given IV
  Other Names: AKR1C3-activated Prodrug OBI-3424; AKR1C3-activated Prodrug TH-3424; Aldo-keto Reductase 1c3-activated Prodrug OBI-3424; AST-3424; OBI 3424; OBI-3424; OBI3424; TH 3424; TH-3424; TH3424
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspirate
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography

SUMMARY:
This phase I/II trial studies the safety, side effects and best dose of OBI-3424 and how well it works in treating patients with T-cell acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Chemotherapy drugs, such as OBI-3424, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. OBI-3424 may reduce the amount of leukemia in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of AKR1C3-activated prodrug OBI-3424 (OBI-3424) and to determine the maximum tolerated dose (MTD) of OBI-3424 in this regimen for patients with relapsed/refractory T-cell acute lymphoblastic leukemia (T-ALL)/T-cell lymphoblastic lymphoma (T-LBL). (Phase I) II. To assess the response rate (complete remission [CR] or CR with incomplete count recovery [CRi]) of patients treated with OBI-3424 at the maximum tolerated dose (MTD) determined in the Phase I portion of the trial in this patient population. (Phase II)

SECONDARY OBJECTIVES:

I. To estimate the frequency and severity of toxicities of OBI-3424 in this patient population.

II. To estimate event-free survival (EFS), relapse-free survival (RFS) and overall survival (OS) in this patient population.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To estimate minimal/measurable residual disease (MRD) negativity (among patients who achieve CR or CRi).

II. To assess AKR1C3 expression levels in this patient population. III. To evaluate associations between AKR1C3 expression and response to OBI-3424, achievement of MRD-negative remission, and relapse from remission.

IV. To bank specimens for future research.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive AKR1C3-activated prodrug OBI-3424 intravenously (IV) over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients who have not achieved a partial remission (PR) by the 4th cycle of treatment are removed from the study (unless clinically benefiting in the opinion of the treating investigator). Patients undergo blood sample collection during screening and cerebrospinal fluid (CSF) sample collection on study. Patients also undergo bone marrow aspirate or core biopsy and may undergo computed tomography (CT) scan throughout the study.

After completion of study treatment, patients are followed up every month for 1 year, every 2 months for 1 year, every 3 months for 1 year, and then every 6 months for up to 5 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of relapsed or refractory T-cell acute lymphoblastic leukemia (T-ALL) based on World Health Organization (WHO) classification. Patients with relapsed/refractory T-cell lymphoblastic lymphoma are eligible if lymphoblasts are >= 5% in the bone marrow or in the peripheral blood by morphology or flow cytometry
* Patients must have evidence of acute leukemia in their peripheral blood or bone marrow. Patients must have >= 5% lymphoblasts in the peripheral blood or bone marrow within 14 days prior to registration. Patients with only extramedullary disease are not eligible
* Patients ≥ 18 years of age must be refractory to or have relapsed following a standard induction chemotherapy. Patients < 18 years of age must have relapsed or must be refractory after 2 or more chemotherapy cycles (example: induction and consolidation)

  * A standard chemotherapy induction regimen is defined as any program of treatment that includes:

    * Vincristine and corticosteroids plus at least one more chemotherapy agent
    * Cytarabine and anthracycline, or
    * High dose cytarabine (defined as at least 1 gr/m^2 per individual dose unless adjustments were required for renal/liver function)
* Patients must have no evidence of central nervous system disease within 28 days prior to registration based on cerebrospinal fluid (CSF) studies. Patients with clinical signs or symptoms consistent with central nervous system (CNS) involvement must have a lumbar puncture which is negative for CNS involvement; the lumbar puncture must be completed within 28 days prior to registration. Patients with CNS1 or CNS2 are eligible; however patients with CNS3 are not eligible
* Note that the patients may receive intrathecal chemotherapy with the initial lumbar puncture. This may count as the first dose of intrathecal therapy required as part of the study
* Prior nelarabine therapy is not required. In addition, for patients ≥ 18 years of age who received nelarabine during initial induction or post-remission treatment are eligible only if the physician does not feel they would benefit from other, multi-agent chemotherapy
* Patients must not have had chemotherapy or investigational agents within 14 days prior to registration except for corticosteroids, oral 6-mercaptopurine, oral methotrexate, vincristine, intrathecal chemotherapy, or hydroxyurea. For participants who have received radiation therapy, at least 7 days must have elapsed from the end of radiation prior to registration and participants must not currently be experiencing toxicities from radiation therapy
* Patients must not have undergone allogeneic hematopoietic transplant within 90 days prior to registration
* Patients must have no evidence of active >= grade 2 acute graft versus host disease (GVHD) or moderate or severe limited chronic GVHD. Patients must have no history of extensive GVHD of any severity within 90 days prior to registration. Patients who are post-transplant must be off calcineurin inhibitors for at least 21 days to be eligible. Extensive GVHD is defined as 1) generalized skin involvement or 2) localized skin involvement and/or hepatic dysfunction plus liver histology or cirrhosis or involvement of eye or minor salivary organ or oral mucosa or any other target organ
* Patients must be >= 12 years of age
* Patients ≥ 16 years of age must have a Zubrod Performance Status of 0-3. Patients < 16 years of age must have a Lansky score of ≥ 50
* Patients must not have systemic fungal, bacterial, viral or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment) within 14 days prior to registration
* Patients ≥ 18 years of age must have creatinine clearance > 30 mL/min within 14 days prior to registration according to the Cockcroft Gault equation
* Patients 12-17 years of age must have adequate renal function within 14 days prior to registration defined as serum creatinine ≤ 1.5 x institutional upper limit of normal (ULN) according to age or a calculated estimated glomerular filtration rate (eGFR) (based on Schwartz formula) or radioisotope glomerular filtration rate (GFR) ≥ 50ml/min/1.73 m^2
* Patients must have direct bilirubin =< 1.5 x institutional upper limit of normal (ULN) within 14 days prior to registration
* Patients must have alanine aminotransferase (ALT) =< 3.0 x institutional upper limit of normal (ULN) or =< 5.0 x ULN (if thought to be related to leukemic involvement) within 14 days prior to registration
* Prothrombin time (PT)/partial thromboplastin time (PTT)/ fibrinogen (as clinically indicated for example but not limited to history of bleeding or active bleeding, concern for disseminated intravascular coagulation) (within 14 days prior to registration to obtain baseline measurements)
* From metabolic panel (comprehensive or basic): sodium, potassium, chloride, carbon dioxide (CO2), and blood urea nitrogen (BUN) (within 14 days prior to registration to obtain baseline measurements)
* Patients must be able to safely discontinue use of strong inhibitors/inducers of CYP3A4 or PgP-g-p and must be able to safely discontinue use of naproxen for 48 hours before and after each dose of OBI-3424
* Patients with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test within 6 months prior to registration. (HIV viral load testing is required only for patients with known HIV infection). Patients must not be receiving antiviral therapies that are known strong inhibitors or inducers of CYP3A4
* Patients with evidence of chronic hepatitis B virus (HBV) infection may be eligible provided that they have an undetectable HBV viral load within 28 days prior to registration. Patients may be currently receiving HBV treatment. (HBV viral load testing is required only for patients with known HBV infection). Patients must not be receiving antiviral therapies that are known strong inhibitors or inducers of CYP3A4
* Patients with known history of hepatitis C virus (HCV) infection may be eligible provided that they have an undetectable HCV viral load within in 28 days prior to registration. Patients may be currently receiving treatment. (HCV viral load testing is required only for patients with known HCV infection). Patients must not be receiving antiviral therapies that are known strong inhibitors or inducers of CYP3A4
* Patients must not have a known history of prolonged QT interval by Fridericia (QTcF) (interval > 450 msec for males; > 470 msec for females). Patients that had transient prolongation of QTc secondary to medications or electrolyte abnormalities are not excluded if the QTc normalized and remain within acceptable QTcF range (interval > 450 msec for males; > 470 msec for females). Additionally, suspected medications should be no longer required or used, and electrolyte abnormalities must have normalized
* Patients must not be pregnant or nursing due to the teratogenic potential of the drug used on this study. Females of reproductive potential must have a negative serum pregnancy test within 14 days prior to registration. Women/men of reproductive potential must have agreed to use an effective contraceptive method during and up to 6 months after treatment. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must not have other active malignancies for which they have received treatments within 6 months prior to registration excluding localized malignancies that do not require systemic treatment
* Patients must agree to have bone marrow and blood specimens submitted for MRD testing
* Patients must be offered the opportunity to participate in specimen banking. With patient consent, residuals from specimens submitted will be retained and banked for future research
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with fedral, local, institutional and Central Institutional Review Board (CIRB) guidelines unless they are unable to provide consent based on age (< 18 years) or based on impaired decision-making capabilities. For patients < 18 years of age or with impaired decision making capabilities, parents or other legally authorized representatives must sign and give informed consent on behalf of study participants in accordance with applicable federal, local, institutional and CIRB regulations
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* This trial will use a slot reservation system to enroll the Phase I portion of the study. Patients planning to enroll at this phase of the study must first have a slot reserved in advance of the registration. All site staff will use OPEN to create a slot reservation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase I) | Up to 21 days
  The regimen will be considered safe and the MTD determined if the dose-limiting toxicity rate is < 33%.
Response rate (complete remission [CR] or CR with incomplete count recovery [CRi]) (Phase II) | Up to 5 years

SECONDARY OUTCOMES:
Incidence of adverse events | Up to the time of relapse, assessed up to 5 years
  Toxicities will be captured and described. The probability of any particular toxicity can be estimated to within at most +/- 17% (95% confidence interval).
Overall survival | From the day of registration on study until death from any cause with observations censored on the day of last contact for patients not known to have died, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.
Event-free survival | From the date of initial registration on study until the first of the following events: death from any cause, relapse from remission (CR or CRi) or completion of protocol therapy without documentation of CR or CRi, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.
Relapse-free survival | From the date the patient first achieves CR or CRi until relapse from CR/CRi or death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
Minimal residual disease (MRD) rate | Up to 5 years
  The MRD rate for responders will be reported as a point estimate with an exact binomial confidence interval.
AKR1C3 expression | Up to 5 years
  A post-hoc analysis of AKR1C3 expression is planned.
Association between AKR1C3 and MRD-negative remission (CR or CRi) status | Up to 5 years
  Will analyze all patients treated at the MTD.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali S Advani, Principal Investigator — SWOG Cancer Research Network
Locations (163):
- United States (163):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Valley Medical Center, Renton, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin